CLINICAL TRIAL: NCT05996042
Title: A Randomized Controlled Trial of Time-restricted Diet Combined With Multimodal Aerobic Exercise Intervention on Cardiovascular and Metabolic Health in a Sedentary Population
Brief Title: Time-restricted Diet Combined With Multimodal Aerobic Exercise
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RCT of Sedentary Population
Record Dates: First submitted 2023-04-13; First posted 2023-08-16 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-04

CONDITIONS: Healthy Population
Keywords: Sedentary; Time-restricted diet; Exercise intervention
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Time-restricted diet group (Other): Subjects in this group were given a limited diet every Tuesday, Thursday and Saturday. They were only allowed to eat from 7am to 3pm on the same day, and only allowed to drink purified water during other periods, namely an 8-hour eating window and a 16-hour fasting period
  Interventions: Behavioral: Time-restricted diet
- Multimode aerobics group (Other): Subjects in this group performed multi-mode aerobic exercise from 6:00 PM to 7:00 PM on Monday, Wednesday and Friday under the unified guidance of the physical education teacher of the Health Science Center in the gymnasium and sports field of Peking University Health Science Center, including aerobics, yoga and comprehensive physical training
  Interventions: Behavioral: Time-restricted diet
- A combination of time-restricted diet and multimodal aerobic exercise (Experimental): Subjects in this group received the same time-limited dietary intervention every Tuesday, Thursday and Saturday according to the above requirements of the single time-limited dietary group, and the same multi-mode aerobic exercise intervention every Monday, Wednesday and Friday according to the above requirements of the single multi-mode aerobic exercise group.
  Interventions: Behavioral: Time-restricted diet

INTERVENTIONS:
Behavioral: Time-restricted diet — On Tuesdays, Thursdays and Saturdays, only eating is allowed between 7am and 3pm. The rest of the time, only drinking pure water is allowed, which is an eight-hour eating window and a 16-hour fasting period.
  On Mondays, Wednesdays and Fridays, under the unified guidance of the physical education teachers of the Health Science Department from 6:00 PM to 7:00 PM, the venue is the gymnasium and sports field of Peking University Health Science Center. The exercise items include aerobics, yoga and comprehensive physical training.
  Other Names: Multimodal aerobic exercise

SUMMARY:
Objective: This study aims to compare the effects of a combination of time-restricted diet and multimodal aerobic exercise (calisthenics, yoga, and comprehensive physical training) on cardiovascular and metabolic health in a sedentary population with both interventions alone.

Study design. Randomized controlled trial Participants: Sedentary (average sitting time greater than 6 hours per day over the past six months, and average moderate-intensity physical activity less than 125 minutes per week or vigorous-intensity physical activity less than 75 minutes per week as assessed by the International Physical Activity Questionnaire).

Sample size: 81 Study grouping and intervention measures: Subjects who signed informed consent and met the inclusion/exclusion conditions were randomly divided into the following three groups according to gender stratification, with 27 participants in each group: single time-limited diet group, single multi-mode aerobic exercise (aerobics, yoga and comprehensive physical training) group, and combination of time-limited diet and multi-mode aerobic exercise group. The subjects who received the time-restricted diet intervention were allowed to eat only from 7am to 3pm on Tuesdays, Thursdays and Saturdays, and were allowed to drink pure water only during the rest of the day. The subjects who received the multi-mode aerobic exercise intervention carried out the exercise intervention from 6:00 PM to 7:00 PM on Monday, Wednesday and Friday under the unified guidance of the physical education teacher of the Medical Department. All subjects did not limit their total daily energy intake. The intervention lasted eight weeks.

Outcome evaluation indicators: The main indicators of this study were body composition (body fat, muscle mass, fat-free weight, body weight, BMI, body fat percentage, total body water, protein, inorganic salts, limb muscle and extracellular water ratio).

DETAILED DESCRIPTION:
Subjects who signed the informed consent and met the inclusion criteria were randomly divided into the following three groups according to gender stratification:

1. Single time-limited diet group: Subjects in this group were given a time-limited diet every Tuesday, Thursday and Saturday. They were only allowed to eat from 7am to 3pm on the same day, and only allowed to drink purified water during other periods, namely an 8-hour eating window and a 16-hour fasting period. Total daily energy intake is not restricted, and food selection is recommended in accordance with the Dietary Guidelines for Chinese Residents (2022). Subjects in this group were required to maintain the original physical activity frequency;
2. Independent multi-mode aerobic exercise group: Subjects in this group will do multi-mode aerobic exercise from 6:00 PM to 7:00 PM on Mondays, Wednesdays and Fridays under the unified guidance of the physical education teacher of the Health Science Department (see Attachment 3 for details). The venue is the gymnasium and sports ground of Peking University Health Science Center, and the exercise items include aerobics, yoga and comprehensive physical training, see attachment for details. Subjects in this group do not limit their daily total energy intake, and it is recommended to choose food according to the Dietary Guidelines for Chinese Residents (2022).
3. Combined group of time-limited diet and multi-mode aerobic exercise: Subjects in this group received the same time-limited diet intervention according to the above requirements of the single-mode diet group every Tuesday, Thursday and Saturday, and the same multi-mode aerobic exercise intervention according to the above requirements of the single-mode aerobic exercise group every Monday, Wednesday and Friday. Total daily energy intake is not restricted, and food selection is recommended in accordance with the Dietary Guidelines for Chinese Residents (2022).

ELIGIBILITY:
Inclusion Criteria:

1. In the past six months, the average daily sitting time was more than 6 hours, and the average weekly moderate-intensity physical activity time was less than 125 minutes or high-intensity physical activity time was less than 75 minutes as assessed by the International Physical Activity Questionnaire (JAMA Intern Med. 2022 Jun 1; 182(6):650-659, J Sport Health Sci. 2022 Mar; 11(2): 164 -- 171. And Global recommendations on physical activity for health);
2. BMI of 18.5-30 kg/m 2, age 18-50, where BMI= weight (kg)/height 2 (m);
3. Weight change less than 3 kg in the last six months;
4. Unlimited hours or other types of fasting, such as alternate-day fasting or simulated fasting diets;
5. No cardiovascular metabolic diseases such as hypertension, type 2 diabetes, chronic kidney disease, coronary heart disease and stroke;
6. No movement disorder related diseases, no sports injury history in the past six months.

Exclusion Criteria:

1. Weigh more than 100 kg;
2. Used weight-loss drugs or dietary supplements and used hormone drugs in the past six months;
3. Abnormal liver and kidney function was found by laboratory examination;
4. Women who are pregnant, lactating or planning to become pregnant in the near future;
5. Still unable to skillfully use smart phones and sports bracelets after training;
6. Other circumstances deemed unsuitable for participation in the study by the researchers

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 81 (Estimated)
Dates: Start 2023-08-20 (Estimated); Primary Completion 2023-09-20 (Estimated); Study Completion 2023-10-20 (Estimated)

PRIMARY OUTCOMES:
Body fat | Baseline survey
  Measurements were made using the Inbody 770, using the bioresistive method
Muscle mass | Baseline survey
  Measurements were made using the Inbody 770, using the bioresistive method
Fat-free weight | Baseline survey
  Measurements were made using the Inbody 770, using the bioresistive method
body weight | Baseline survey
  Measurements were made using the Inbody 770, using the bioresistive method in Kg
body weight | 8 weeks after baseline survey
  Measurements were made using the Inbody 770, using the bioresistive method in Kg
Body fat percentage | Baseline survey
  Measurements were made using the Inbody 770, using the bioresistive method in %
Body fat percentage | 8 weeks after baseline survey
  Measurements were made using the Inbody 770, using the bioresistive method in %
Body water | Baseline survey
  Measurements were made using the Inbody 770, using the bioresistive method
Body water | 8 weeks after baseline survey
  Measurements were made using the Inbody 770, using the bioresistive method
Muscle mass | 8 weeks after baseline survey
  Measurements were made using the Inbody 770, using the bioresistive method
Body fat | 8 weeks after baseline survey
  Measurements were made using the Inbody 770, using the bioresistive method
Fat-free weight | 8 weeks after baseline survey
  Measurements were made using the Inbody 770, using the bioresistive method
Body mass index | Baseline survey
  Measurements were made using the Inbody 770, measured by weight(Kg) divided by height(meter) squared
Body mass index | 8 weeks after baseline survey
  Measurements were made using the Inbody 770, measured by weight(Kg) divided by height(meter) squared

SECONDARY OUTCOMES:
Waist circumference | Baseline survey
  The measurements are made by a professional using a tape measure
Waist circumference | 8 weeks after baseline survey
  The measurements are made by a professional using a tape measure
Hip circumference | Baseline survey
  The measurements are made by a professional using a tape measure
Hip circumference | 8 weeks after baseline survey
  The measurements are made by a professional using a tape measure
Blood pressure | Baseline survey
  The measurement was carried out using an electronic sphygmomanometer, and the average value was measured three times in the resting state
Blood pressure | 8 weeks after baseline survey
  The measurement was carried out using an electronic sphygmomanometer, and the average value was measured three times in the resting state
Heart rate | Baseline survey
  The heart rate band was used for measurement, and the resting state was measured three times to take the average value
Heart rate | 8 weeks after baseline survey
  The heart rate band was used for measurement, and the resting state was measured three times to take the average value
Blood Lipid | Baseline survey
  Fasting blood lipid (TC, TG, HDL-C, LDL-C),Blood is drawn by a trained nurse and blood biochemical tests are performed
Blood Lipid | 8 weeks after baseline survey
  Including TC, TG, HDL-C, LDL-C ,blood is drawn by a trained nurse and blood biochemical tests are performed
urine routine | Baseline survey
  Including urinary protein, urinary creatinine, urine collection was followed by routine urine testing at the hospital
urine routine | 8 weeks after baseline survey
  Including urinary protein, urinary creatinine, urine collection was followed by routine urine testing at the hospital
Questionnaire survey | Baseline survey
  Demographic characteristics questionnaire, 4-day 24-hour dietary review, international physical activity questionnaire, sleep quality questionnaire, CNAQ appetite questionnaire
Questionnaire survey | 8 weeks after baseline survey
  Demographic characteristics questionnaire, 4-day 24-hour dietary review, international physical activity questionnaire, sleep quality questionnaire, CNAQ appetite questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Qihuang Gong, Dr, Study Chair — Peking University

IPD SHARING:
Plan to Share IPD: Yes
The anonymous data is then shared with relevant collaborators
Supporting Information: Study Protocol, ICF, CSR, Analytic Code
Time Frame: After the data is anonymized
Access Criteria: Need to reach an agreement and sign a collaboration agreement with the researcher